CLINICAL TRIAL: NCT00476619
Title: Erythropoietin in Radiocontrast Induced Nephropathy (ERIN) Trial
Acronym: ERIN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The exclusion criteria were stringent and enrollment was slow.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Responsible Party: Dr Ajay K Singh, MD MBA FRCP, Brigham and Womens Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2004P000510
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast; Nephropathy; acute renal failure; Erythropoietin; CT scan
MeSH Terms: conditions — Kidney Diseases; Acute Kidney Injury | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erythropoeitin (Placebo Comparator): Subjects will receive a one-time dose of either placebo, or EPO 40,000 U intravenously 30 to 240 minutes prior to intravenous contrast administration.
  Interventions: Drug: erythropoeitin

INTERVENTIONS:
Drug: erythropoeitin — Subjects will receive a one-time dose of either placebo, or EPO 40,000 U intravenously 30 to 240 minutes prior to intravenous contrast administration.
  Other Names: PROCRIT

SUMMARY:
Full Title: A Randomized Controlled Trial of Procrit for the Prevention of Acute Renal Failure in Patients Receiving Intravenous Contrast

Primary Objective: To evaluate the efficacy of a one-time dose of intravenous erythropoietin administration in the prevention or attenuation of contrast-induced acute renal failure.

Secondary Objectives: To evaluate serum and urinary markers of renal injury, including KIM-1, BMP-7, and TGF-b, along with other biomarkers, in subjects receiving intravenous contrast and correlate their expression with clinical outcomes

Study Design: Prospective, multi-centered, randomized, double blind, placebo controlled trial of a one-time dose of EPO. Subjects will be followed for seven days or until hospital discharge, whichever is longer. Total estimated study duration 3 years.

DETAILED DESCRIPTION:
Adult subjects with or without diabetes mellitus Eligibility Criteria: undergoing intravenous contrast administration for computerized axial tomography (CAT Scan) as inpatients.

Subjects will be excluded if they have end-stage renal disease (on dialysis or peritoneal dialysis); any known history of acute renal failure; have hemoglobin ³ 12.0 g/dL; history of use of erythropoietin replacement or transfusion within the prior 3 days; use Glucophage/Metformin or Glucovance; are unable to give their written informed consent; have hemodynamic instability; have uncontrolled hypertension; have any history of current malignancy, where current malignancy is defined as subjects undergoing treatment with chemotherapy or radiation therapy, subjects with known metastatic disease, and those with terminal malignant disease; any history of MI, CVA, active angina or unstable angina within the past three months ; are pregnant or lactating; allergic to intravenous contrast, iodine, erythropoietin, mammalian-cell derived products, or human albumin; patients with seizure disorders or have CT scan done as hospital outpatients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 and over and of either gender.
2. Scheduled to receive CT scan with intravenous contrast dye.
3. Non diabetics or subjects with type 1 or 2 diabetes mellitus
4. Written informed consent.
5. Subjects who are on diuretics and non-steroidal inflammatory agents will not be excluded.
6. Subjects who have received n-acetylcysteine or sodium bicarbonate pre CT scan will not be excluded

Exclusion Criteria:

1. Pregnant or lactating women.
2. End-stage renal disease (on hemodialysis or peritoneal dialysis)
3. A known history of acute renal failure
4. Subjects receiving glucophage/metformin or glucovance
5. Subjects who cannot give written informed consent.
6. Subjects receiving peritoneal dialysis or hemodialysis.
7. Subjects enrolled in another investigational drug study ≤ 30 days of enrollment into the present study.
8. Subjects with a known hypersensitivity or anaphylaxis to contrast dye or iodine.
9. Subjects with known hypersensitivity or anaphylaxis to erythropoietin, mammalian-cell derived products, or human albumin.
10. Age < 18 years
11. Use of any erythropoietin replacement or transfusion within the prior 3 days
12. Baseline Hemoglobin > 12.0 g/dL
13. Uncontrolled hypertension, systolic BP > 180 mmHg or diastolic BP > 110 mmHg in any recording in the past 24 hours.
14. Evidence of hemodynamic instability
15. Subject unable to follow protocol due to mental incompetence or other reason
16. Inaccessibility of medical record
17. Subjects with a history of MI, CVA, active angina or unstable angina within the past three months
18. Subjects with a history of current malignancy, where current malignancy is defined as subjects undergoing treatment with chemotherapy or radiation therapy, subjects with known metastatic disease, and those with terminal malignant disease.
19. Subject with any known history of seizure disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-09; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Comparison of incidence of rise in serum creatinine of 25% or more in the study group vs. placebo | 7 days

SECONDARY OUTCOMES:
Doubling of serum creatinine 2) Need for dialytic support 3) Patient death 4) Comparison of urinary markers of renal injury in subjects in study group vs. placebo and in subjects with and without ARF | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Singh, M.D., Principal Investigator — Brigham and Womens Hospital and Harvard Medical School
Locations (1):
- Brigham and Womens hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879